CLINICAL TRIAL: NCT03991637
Title: Remote Sensing Comprehensive Metabolic Panel
Brief Title: Non-Invasive Blood Test Cross-Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Allen Jr. (Industry)
Collaborators: University of North Dakota (Other)
Responsible Party: Sponsor-Investigator, Joseph Allen Jr., Chief Executive Officer/Biomedical Engineer, Concord Medical Technology Corporation
Organization: Concord Medical Technology Corporation (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-201807-004
Record Dates: First submitted 2019-06-01; First posted 2019-06-19 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Reproducibility of Results; Safety Issues

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NICMP Spectral Reading (Experimental): Non-invasive spectral data is collected from this arm to function as the intervention of interest.
  Interventions: Device: Non-Invasive Comprehensive Metabolic Panel
- Venipuncture CMP (Active Comparator): A standard CMP blood draw is performed to function as the "gold standard" reference value.
  Specifically, the outcome of the experimental arm is cross-validated against the active comparator arm to determine the NICMP accuracy, relative to the venipuncture method.
  Interventions: Device: Non-Invasive Comprehensive Metabolic Panel

INTERVENTIONS:
Device: Non-Invasive Comprehensive Metabolic Panel — The device utilizes spectroscopy and machine learning to detect metabolic analyte concentrations.

SUMMARY:
The study considers a cross-validation approach to determine the effectiveness of a non-invasive comprehensive metabolic panel (NICMP), relative to the venipuncture method. The NICMP machine learned powered device utilizes a light sensor to capture readings from either palm. The study (n=90) proves an agreement and strong correlation with respect to the NICMP and venipuncture blood draw.

ELIGIBILITY:
Inclusion Criteria:

* Undiagnosed population

Exclusion Criteria:

* Diagnosed population, pregnant women, mental heath/disabled, prisoners, fetus or deceased

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Performance of Non-Invasive Comprehensive Metabolic Panel | 2-minutes
  Determine the effectiveness, in terms of accuracy, of the NICMP against the venipuncture CMP (i.e. reference value).

CONTACTS AND LOCATIONS:
Locations (1):
- Altru Health System, Grand Forks, North Dakota, United States